CLINICAL TRIAL: NCT06042309
Title: Improving the Diagnosis and Prevention of Contact Allergy to Rubber Accelerators
Brief Title: Contact Allergy to Rubber Accelerators - a Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Allergy Research Center, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-22058515
Record Dates: First submitted 2023-09-01; First posted 2023-09-18 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Contact Allergy
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: The participants are assigned to either the SLS-group or NON-SLS-group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The forearm randomized to SLS and the order in which the different concentrations of thiurams and carbamates and the control solution are applied to the skin, will be blinded for the reader of the skin reactions and the latter also for the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NON-SLS, Allergic participants (Experimental): Participants allergic to thiurams or carbamates assigned to the NON-SLS group.
  Interventions: Other: Rubber accelerators and control chamber/solution for NON-SLS group; Other: Patch test on back
- NON-SLS, Control participants (Experimental): Participants not allergic to thiurams or carbamates assigned to the NON-SLS group.
  Interventions: Other: Rubber accelerators and control chamber/solution for NON-SLS group; Other: Patch test on back
- SLS, Allergic participants (Experimental): Participants allergic to thiurams or carbamates assigned to the SLS group.
  Interventions: Other: SLS; Other: Rubber accelerators and control chamber/solution for SLS group; Other: Patch test on back
- SLS, Control participants (Experimental): Participants not allergic to thiurams or carbamates assigned to the SLS group.
  Interventions: Other: SLS; Other: Rubber accelerators and control chamber/solution for SLS group; Other: Patch test on back

INTERVENTIONS:
Other: Rubber accelerators and control chamber/solution for NON-SLS group — Repeated exposure to rubber accelerators and control chamber/solution on arms. Three different concentrations of rubber accelerators and one control chamber/solution will be applied on the arms.
  Arms: NON-SLS, Allergic participants; NON-SLS, Control participants
Other: SLS — Exposure to SLS on a randomized arm
  Arms: SLS, Allergic participants; SLS, Control participants
Other: Rubber accelerators and control chamber/solution for SLS group — Repeated exposure to rubber accelerators and control chamber/solution on arms. Two different concentrations of rubber accelerators and one control chamber/solution will be applied on both arms.
  Arms: SLS, Allergic participants; SLS, Control participants
Other: Patch test on back — Patch test on the back with thiurams or carbamates in different concentrations and a control chamber/solution

SUMMARY:
This study will investigate what concentrations of the most common thiurams and carbamates that elicit allergic contact dermatitis under patch test and what concentrations of the rubber accelerators that elicit allergic contact dermatitis by repeated exposures under simulated use conditions. Further, it will investigate whether a damaged skin barrier as caused by wet work increase the severity of the allergic contact dermatitis.

The participants will be assigned to either the SLS (sodium lauryl sulfate)-group or non SLS-group. For the participants of the SLS-group, one volar forearm will be randomized to be pre-irritated with a soap i.e. detergent: sodium lauryl sulfate (SLS) for 24 hours to simulate wet work. The participants of the non SLS-group will not be pre-irritated with SLS.

Following this, the participants' volar forearms will be exposed to thiurams or carbamates and a control solution every night for 7 nights to simulate the repeated exposure to rubber gloves with accelerators. The skin reactions will be read cf. current international guidelines and further quantified using laser Doppler flowmetry.

During the study, all participants will be patch tested on the upper back with rubber accelerators to investigate their current degree of sensitization and the dose-response relationships.

ELIGIBILITY:
Allergic participants

Inclusion Criteria:

* Adults ≥18 years old
* Sensitized to thiurams, carbamates or both.
* Received written and oral information about the study.
* Signed written consent form

Exclusion Criteria:

* Dermatitis on back or arms
* Tattoos or significant scar tissue on exposure areas
* Pregnancy
* Breast feeding
* Recently given birth
* Treatment with systemic immunomodulators within the last 4 weeks
* Treatment with local immunomodulators on arms or back within the last 4 weeks
* Excessive ultraviolet light on arms or back within the last 4 weeks

Healthy Controls:

Inclusion Criteria:

* adults ≥18 years old
* Received written and oral information about the study.
* Signed written consent form

Exclusion Criteria:

* Sensitized to thiurams, carbamates or both.
* Occupational or domestical use of rubber gloves.
* History of atopic dermatitis or contact dermatitis
* Dermatitis on back or arms
* Tattoos or significant scar tissue on exposure areas
* Pregnancy
* Breast feeding
* Recently given birth
* Treatment with systemic immunomodulators within the last 4 weeks
* Treatment with local immunomodulators on arms or back within the last 4 weeks
* Excessive ultraviolet light on arms or back within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Reading of skin reactions | Day 0, Day 1 (only participants' arms in the SLS-group), Day 2 and Day 3 or Day 4, and Day 7, and Day 8. Further, eventually, if any reactions occur up to Day 16.
  Development of dermatitis by reading of skin reactions based on international dermatitis scoring guidelines.
Skin blood flow | Day 0, Day 1 (only participants' arms in the SLS-group), Day 2 and Day 3 or Day 4, and Day 7, and Day 8. Further, eventually, if any reactions occur up to Day 16.
  Changes in blood flow on the arms using laser doppler flowmetry

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Dermatology, Gentofte Hospital, Videncenter For Allergi, Hellerup
  - Department of Dermatology and Allergy, Odense University Hospital (OUH), Odense

REFERENCES:
- [Derived] Kursawe Larsen C, Johansen JD, Zachariae C, Svedman C, Bergendorff O, Mortz CG, Schwensen JFB. Thresholds for Contact Allergy to a Rubber Accelerator: TETD-Determined by Serial Dilution Patch Testing and a Simulated Glove-Use Model. Contact Dermatitis. 2025 Aug;93(2):138-147. doi: 10.1111/cod.14817. Epub 2025 May 16. PMID 40375756